CLINICAL TRIAL: NCT02341040
Title: Evaluation of Potential Allergenicity of New Wheat Varieties
Status: Terminated | Type: Observational
Why Stopped: insufficient subjects recruited in allotted time
Sponsor: University of Colorado, Denver (Other)
Collaborators: Monsanto Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-1416; UL1TR001082 (NIH)
Record Dates: First submitted 2015-01-06; First posted 2015-01-19 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Food Allergy; Wheat Allergy
Keywords: wheat allergy; food allergy; pediatric
MeSH Terms: conditions — Food Hypersensitivity; Wheat Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subjects may opt to have extra blood drawn. This sample will be de-identified and sent to the sponsor, Monsanto, for future study that is yet to be determined.
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is to determine accurate blood test levels that can predict whether or not subjects are truly allergic to certain foods. In this study, subjects that are clinically documented to be wheat-allergic will participate in a double blind oral food challenge. Blood will be collected from the subject to evaluate the potential allergenicity of proteins introduced into genetically modified crops and evaluate wheat-specific immunoglobulin-e (IgE) antibody reactivity to biotech and conventional wheat varieties.

DETAILED DESCRIPTION:
The prevalence of food allergy is increasing in the pediatric population. A diagnosis of food allergy carries significant medical, nutritional, and psychological implications for both patients and their families. Therefore, making an accurate diagnosis is critical. However, the diagnosis of symptomatic food allergy continues to be a challenge for allergists and other practicing physicians. The patient's clinical history remains a key component in diagnosing food allergy. Skin prick testing and food-specific immunoglobulin-e (IgE) testing act as secondary tools to aid in the evaluation process, but these tests also suffer from a high rate of false positivity. For specific IgE levels below the cutoffs to these foods, however, supervised oral food challenges (OFCs) may be necessary to establish the diagnosis of symptomatic food allergy, as the sensitivity of these values is relatively low. Currently, the double-blind, placebo-controlled food challenge (DBPCFC) remains the gold standard for the diagnosis of food allergy. OFCs have their own inherent drawbacks: they are not always readily available to all patients, they are time-consuming, and they are potentially dangerous due to their risk of anaphylaxis.

Wheat is one of the eight allergenic foods that are responsible for approximately 90% of all food allergies. Wheat is less allergenic than other foods in this group and less likely to cause multi-organ, severe, life-threatening reactions. Allergy to wheat is more prevalent in children than adults and is considered a transient allergy of infancy/childhood. Wheat allergy is often outgrown in early childhood, in most cases by age 3-5 years, but 35% show a persistent allergy into adolescence. While previous studies using food-specific IgE antibodies have determined diagnostic decision points that indicate a high likelihood of clinical reactivity for certain foods, namely milk, egg, peanut, and fish, wheat-specific IgE levels do not seem to be useful predictors of food challenge outcome, enabling reduction in need for food challenges. Furthermore, false-positive IgE reactions to wheat and other cereals are frequently seen in grass-allergic patients due to insignificant cross-reactivity between water/salt-soluble proteins. Therefore, identification of wheat proteins associated with symptoms to wheat is of importance.

Gliadins in particular have been implicated in allergy to wheat, both in IgE-mediatedallergy and the non-IgE mediated celiac allergy. IgE antibodies to ω-5-gliadin have been found in children with immediate reactions to ingested wheat, and published results show that increased levels of IgE to ω-5-gliadin correlate with the outcome of food challenges. In a Finnish study, all children with IgE antibodies to ω-5-gliadin reacted with immediate symptoms to wheat challenges, while all patients with delayed or negative challenge test results showed no detectable IgE antibodies to ω-5-gliadin.15 In a Japanese cohort, the presence of elevated ω-5-gliadin-specific IgE antibodies was associated with immediate symptoms with wheat food challenges and also in patients with a strong convincing history of wheat allergy who were not challenged due to risk of anaphylaxis. Furthermore, patients with severe reactions upon challenge had significantly higher levels of ω-5-gliadin-specific IgE antibodies compared to children with mild or moderate symptoms. In a multicenter Japanese study, Ebisawa et al. showed a significant relationship between the probability of wheat allergy and the concentration of ω-5-gliadin-specific IgE antibodies with 2.6-fold increased risk. In a study of mixed German and American subjects, ω-5-gliadin-specific IgE antibodies did not correlate with food challenge outcomes in patients with suspected allergy. However, the sample size in this study was much smaller than in others, and the German population included more patients with non-IgE mediated wheat allergy with delayed symptoms, almost half of the German cohort. Nonetheless, ω-5-gliadin-specific IgE antibodies may differ among populations in Asia, Europe, and the United States due to dietary habits and genetics, and further study is warranted, especially in a larger U.S. cohort.

Food crops that have been developed through agricultural biotechnology for commercial use are thoroughly assessed for their safety. One of the key elements in the safety assessment of a genetically improved crop is an evaluation of potential changes in their allergenic properties. Allergenic properties of the crop can potentially be altered if a known allergen or a protein that has high potential to become an allergen is introduced. In addition, the level of expression of endogenous allergens might be altered as a result of transformation and insertion of the new gene into the plant genome.

Since wheat is a known allergenic food crop, international guidelines require analyses to determine if the introduction of the genes and production of the recombinant proteins in wheat cause an unintended change in the levels of endogenous allergenic proteins. To address this question, levels of wheat-specific IgE binding observed in the biotechnology derived wheat varieties are compared to the set of binding values observed in reference wheat varieties that are already on the market. Determining the levels of direct IgE binding using an enzyme linked immuno-sorbent assay (ELISA) has been shown to be an appropriate method to perform such comparisons, especially when the assay is validated and calibrated prior to the production of data. This comparison is important as it will enable determinations of whether there is heterogeneity in wheat-allergic patients with wheat allergy in terms of a predominant trigger. Ultimately, crops may be engineered to eliminate culprit components if predominant.

Food challenge outcomes and standard ImmunoCAP IgE assays to wheat will be compared to CRD wheat testing in this study (Thermo Fisher Scientific, Waltham, MA). When evaluated together with clinical history, skin test reactivity, and OFC outcomes, responses to individual components may be able be used to predict food challenge responsiveness. With respect to intact wheat-specific IgE levels, in two previous studies using these, a true 95% positive predictive value cutoff to predict reactivity at OFC could not be determined to wheat, although a physician challenge was suggested at an estimated wheat level of 26 kU/L to determine possible reactivity.6,7 However, these studies are now over a decade old and pre-dated component resolved diagnostics (CRD). CRD to major proteins ω-5-gliadin may prove to be more beneficial in determining predictive levels of IgE and positive OFC outcomes to wheat. Therefore, in addition to determining wheat component patterns that could predict OFC outcomes, the investigators hope to determine 95% predictive decision points for each of the individual components and compare these to the decision points estimated by the ImmunoCAP assay to wheat.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 year to 21 years of any sex and any race
* Physician-diagnosed food allergy to wheat with convincing clinical history of food allergy to wheat AND a skin prick test positive to wheat (diameter of wheal 3 mm or greater than negative control) or a detectable serum food-specific IgE level (ImmunoCAP > 0.35 kUA/L) to wheat within the previous 12 months or at the time of entry into the study
* If no history of clinical reactivity to wheat, then a positive skin prick test to wheat (diameter of wheal 3 mm or greater than negative control) OR a detectable serum food-specific IgE level to wheat within the previous 12 months or at the time of entry into the study
* Patients who meet any of the following criteria are eligible for enrollment as study participants if they meet all other criteria, but will not undergo a DBPCFC:

  * Recent (within one year) failed open OFC
  * Positive DBPCFC to wheat at CHCO
  * Recent (within one year) exposure to wheat resulting in immediate IgE-mediated allergic symptoms (within 2 hours of ingestion; symptoms such as urticaria, angioedema, congestion, rhinorrhea, wheezing, respiratory compromise, hypoxia, hypotension)
* Written informed consent from parent/guardian and assent (when age appropriate).
* Willingness to submit specimen for laboratory serum IgE testing
* Willingness to submit lab specimen for ELISA testing

Exclusion Criteria:

* Inability to discontinue antihistamines for skin prick testing and OFCs
* FEV1 value <80% predicted OR any clinical features of moderate or severe persistent asthma, as defined by the 2007 NHLBI guidelines table for classifying asthma, at the time of entry into the study
* Use of >500 μg/day fluticasone or equivalent
* Asthma requiring either:

  * 1 hospitalization in the past year for asthma, or
  * 1 ER visit in the past 6 months for asthma
* Use of steroid medications (IV, IM or oral) for asthma in the following manners:

  * history of daily oral steroid dosing for >1 month during the past year, or
  * steroid course/burst in the past 3 months (except for steroid dosing used in the treatment of an allergic reaction during the DBPCFC), or
  * 2 steroid courses/bursts in the past year.
* History of intubation due to allergies or asthma
* Diagnosis of active eosinophilic gastrointestinal disease in the past year
* Severe atopic dermatitis, as assessed by a Three-Item Severity Score of 6 or greater

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric and adult subjects between the ages of 1 (inclusive) to 21 years (inclusive) that have sensitivity to wheat
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Determine the relationship between whole wheat-specific IgE and IgE to components | ~2 weeks
  Logistic regression analyses will be performed to establish diagnostic decision pointsindicating a high likelihood of symptomatic food allergy to wheat, thus potentiallypreventing unnecessary food challenges for patients with wheat allergy..

SECONDARY OUTCOMES:
Determine the relationship between IgE components and oral food challenge | ~2 weeks
  The investigators will evaluate IgE to components Tri a 14, Tri a 19, and Tri a Aa_TI, and Oral Food Challenges outcomes.
Determine the Cross-Reactivity between wheat and grass allergens | ~1 month
  To assess cross-reactivity between wheat and grass allergens in wheat-allergic patients.
Determine the Potential Allergenicity | ~1 month
  To evaluate the potential allergenicity of putative wheat allergens.
Establish a Serum Repository | ~2 weeks
  To establish a serum repository at Monsanto of wheat-reactive allergic patients.

CONTACTS AND LOCATIONS:
Overall Officials: David Fleischer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States